CLINICAL TRIAL: NCT02259751
Title: A Phase I, Randomised, Double-blind, Placebo-controlled Study to Determine Pharmacodynamic Effects and Pharmacokinetics of a Single Oral Dose of 320 mg KUC 7483 CL in Patients With Spinal Cord Injury and Neurogenic Detrusor Overactivity
Brief Title: Study to Determine Pharmacodynamic Effects and Pharmacokinetics of KUC 7483 CL in Patients With Spinal Cord Injury and Neurogenic Detrusor Overactivity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1207.4
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

ARMS (2):
- KUC 7483 CL (Experimental)
  Interventions: Drug: KUC 7483 CL
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KUC 7483 CL
  Arms: KUC 7483 CL
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to investigate pharmacodynamic effects and pharmacokinetics of KUC 7483

ELIGIBILITY:
Inclusion Criteria:

1. Male patients with acquired suprasacral spinal cord injury practicing intermittent catheterization under stable condition as determined by the investigator
2. Recovery from spinal shock in posttraumatic patients
3. Aged 18 - 70 years
4. BMI range ≥ 18.5 and < 29.9 kg/m2
5. Documented neurogenic detrusor overactivity as shown by urodynamics within the last 12 months prior to study start and confirmation by the baseline urodynamics (day 2). Detrusor overactivity is defined as a non-volitional increase in detrusor pressure of > 6 cm H2O. Detrusor sphincter dyssynergia may be facultative
6. Written informed consent consistent with International committee on harmonization (ICH)/ Good Clinical Practice (GCP) and local legislation given prior to any study procedures
7. Ability and willingness to comply with study treatment regimen and to attend study

Exclusion Criteria:

1. A total daily volume of urine > 3000 ml as verified in the micturition diary before randomization
2. Treatment with drugs with known anticholinergic effect on the detrusor and/or alpha-blockers, 7 days prior to inclusion visit 2
3. Treatment with botulinus toxin, capsaicin or resiniferatoxin in the last 6 months prior to the study
4. Unstable dosage of any drug or the expectation of initiation of such a treatment during the trial
5. Use of agonists or antagonists at beta-adrenoceptors (The following drugs may nevertheless be used since they do not act upon beta-3 adrenoceptors in therapeutic doses: atenolol, bisoprolol, carvedilol, metoprolol, propranolol, salbutamol and salmeterol)
6. Neurological diseases other than suprasacral spinal cord injury, affecting urinary bladder function
7. Significant stress incontinence as determined by the investigator
8. Non-functional bladder outlet obstruction as determined by the investigator
9. Dilatation of the upper urinary tract
10. Low compliance bladder (Compliance < 20 mL/cm H2O)
11. Detrusor hyporeflexia/areflexia and bradykinesia/tremor of the external urethral sphincter
12. Prostatic or bladder carcinoma
13. Acute urinary tract infection during the run-in period or during study period
14. History of interstitial cystitis
15. Surgery of the prostate, the urinary bladder, the urethra, and thermotherapy, ultrasound or laser therapy of the prostate for 12 months prior to enrolment to the study
16. Pelvic radiation therapy
17. Use of indwelling catheter
18. Any electro stimulation therapy within the 14 days prior to inclusion visit 2
19. Significant hepatic or renal disease defined as twice the upper limit of the reference range, regarding serum concentrations of Aspartate transaminase ((SGOT) (AST)), Alanine transaminase ((SGPT) ALT)), Alkaline phosphatase (ALP), and/or creatinine > 1.4 mg/dl
20. Diseases or any condition, in which treatment with ß3-adrenoceptors agonists is contraindicated
21. Participation in another clinical trail 8 weeks preceding to enrolment in this study or during study period
22. Patients with any severe medical or any other condition which in the opinion of the investigator makes the patient unsuitable for inclusion
23. Allergic to KUC-7483 or its excipients
24. Patients with Diabetes mellitus type 1 or 2 treated with oral antidiabetic drugs or insulin (any formulation)

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2004-02; Primary Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in "volume at first contraction" | 2 hours post dosing
Change from baseline in "volume at first contraction" | 6 hours post dosing

SECONDARY OUTCOMES:
Change from baseline in Detrusor pressure at first contraction | 2 and 6 hours post dosing
Change from baseline in Maximum amplitude of involuntary detrusor contraction | 2 and 6 hours post dosing
Change from baseline in Volume at first incontinence episode | 2 and 6 hours post dosing
Change from baseline in compliance | 2 and 6 hours post dosing
Change from baseline in Maximum cystometric capacity | 2 and 6 hours post dosing
Change from baseline in Detrusor pressure at maximum flow induced by triggering | 2 and 6 hours post dosing
Change from baseline in Post-triggering residual urinary volume | 2 and 6 hours post dosing
AUC0-∞ (area under the concentration time curve of KUC 7322 ZW in plasma over the time interval from 0 extrapolated to infinity) | up to 24 hours post dosing
Cmax (maximum concentration of KUC 7322 ZW in plasma) | up to 24 hours post dosing
AUC0-tz (area under the concentration-time curve of KUC 7322 ZW in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 24 hours post dosing
AUC0-24 (Area under the concentration time curve of KUC 7322 ZW in plasma over the time interval 0 to 24 hours) | up to 24 hours post dosing
tmax (time from dosing to the maximum concentration of KUC 7322 ZW in plasma) | up to 24 hours post dosing
λz (terminal rate constant of KUC 7322 ZW in plasma) | up to 24 hours post dosing
t1/2 (terminal half-life of KUC 7322 ZW in plasma) | up to 24 hours post dosing
MRTpo (mean residence time of KUC 7322 ZW in the body after po administration) | up to 24 hours post dosing
CL/F (apparent clearance of KUC 7322 ZW in the plasma after extravascular administration) | up to 24 hours post dosing
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 24 hours post dosing
Aet1-t2 (amount of KUC 7322 ZW that is eliminated in urine from the time interval t1 to t2) | up to 24 hours post dosing
fet1-t2 (fraction of administered drug excreted unchanged in urine from time point t1 to t2) | up to 24 hours post dosing
CLR,t1-t2 (renal clearance of KUC 7322 ZW in plasma from the time point t1 until the time point t2) | up to 24 hours post dosing
Number of patients with adverse events | up to 26 days
Number of patients with clinically significant changes in vital signs | up to 24 hours post dosing
  Blood Pressure
Assessment of tolerability by investigator on a 4-point scale | 10 days post dosing
Assessment of tolerability by patient on a 4-point scale | 10 days post dosing